CLINICAL TRIAL: NCT03703700
Title: The Application of Zishen Yutai Pill in Aged Women Undergoing in Vitro Fertilization-embryo Transfer: a Multi-center Double-blind Randomized Controlled Trial
Brief Title: The Application of Zishen Yutai Pill in Aged Women Undergoing IVF-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Dongzi Yang, professor，Chief Physician，doctoral supervisor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018112704
Record Dates: First submitted 2018-08-05; First posted 2018-10-12 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Infertility, Female
Keywords: IVF-ET; infertility; aged; women
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Zishen Yutai

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zishen Yutai pill group (Experimental): Patients who undergo the long-term protocol will start taking Zishen Yutai Pill on the day of pituitary suppression, 5g three times a day (Stopping on the first 1-4 days of menstruation), and patients who undergo the antagonist protocol will start taking Zishen Yutai Pill on the 19th to 23rd day of the previous menstruation cycle, 5g three times a day (Stopping on the first 1-4 days of menstruation). The drug will be taken till 2 weeks after transplantation. If the test result is confirmed as biochemical pregnancy (HCG>50 IU/L), patients continue to take pills till 3 weeks after the clinical pregnancy determined by the ultrasound. If it is determined that the pregnancy test is negative, stop the drug.
  Interventions: Drug: Zishen Yutai Pill
- Placebo group (Placebo Comparator): Patients who undergo the long-term protocol will start taking Placebo on the day of pituitary suppression, 5g three times a day (Stopping on the first 1-4 days of menstruation), and patients who undergo the antagonist protocol will start taking Placebo on the 19th to 23rd day of the previous menstruation cycle, 5g three times a day (Stopping on the first 1-4 days of menstruation). The drug will be taken till 2 weeks after transplantation. If the test result is confirmed as biochemical pregnancy (HCG>50 IU/L), patients continue to take pills till 3 weeks after the clinical pregnancy determined by the ultrasound. If it is determined that the pregnancy test is negative, stop the drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zishen Yutai Pill — Patients who undergo the long-term protocol will start taking Zishen Yutai Pill on the day of pituitary suppression, 5g three times a day (Stopping on the first 1-4 days of menstruation), and patients who undergo the antagonist protocol will start taking Zishen Yutai Pill on the 19th to 23rd day of the previous menstruation cycle, 5g three times a day (Stopping on the first 1-4 days of menstruation). The drug will be taken till 2 weeks after transplantation. If the test result is confirmed as biochemical pregnancy (HCG>50 IU/L), patients continue to take pills till 3 weeks after the clinical pregnancy determined by the ultrasound. If it is determined that the pregnancy test is negative, stop the drug.
  Arms: Zishen Yutai pill group
Drug: Placebo — Patients who undergo the long-term protocol will start taking Placebo on the day of pituitary suppression, 5g three times a day (Stopping on the first 1-4 days of menstruation), and patients who undergo the antagonist protocol will start taking Placebo on the 19th to 23rd day of the previous menstruation cycle, 5g three times a day (Stopping on the first 1-4 days of menstruation). The drug will be taken till 2 weeks after transplantation. If the test result is confirmed as biochemical pregnancy (HCG>50 IU/L), patients continue to take pills till 3 weeks after the clinical pregnancy determined by the ultrasound. If it is determined that the pregnancy test is negative, stop the drug.
  Arms: Placebo group

SUMMARY:
To explore the application of Zishen Yutai Pill in controlled ovarian stimulation and effect on pregnancy outcome in aged women undergoing in vitro fertilization-embryo transfer.

DETAILED DESCRIPTION:
This will be a multi-center double-blind randomized controlled trial, which aims to explore the application of Zishen Yutai Pill in controlled ovarian stimulation and effect on pregnancy outcome in aged women undergoing in vitro fertilization-embryo transfer.The target population will be infertile women aged between 35 and 42 years, BMI<28kg/m2 and bilateral ovaries who undergo IVF-ET (long or antagonist protocol). Qualified 1,466 patients are randomized into either of two groups.They will be randomized to receive either Zishen Yutai Pill or the placebo. The pregnancy test results and pregnancy complications will be followed up by checking medical records and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* infertile women aged ≥35 and ≤42 years;
* intend to undergo IVF/ICSI-ET (GnRH-a long protocol or GnRH-ant protocol);
* BMI<28kg/m2;
* bilateral ovaries exist;
* patients who voluntarily signed the informed consent and agreed to be followed up as required by the study protocol.

Exclusion Criteria:

* repeated implantation failure (previous three times or more IVF/ICSI-ET failure);
* adenomyosis, uterine line constricted by uterine fibroid;
* untreated bilateral hydrosalpinx;
* endometrial diseases that have not been cured ;
* known diseases that are not suitable for undergoing assisted reproductive technology or at the present not suitable for pregnancy;
* patients who have taken traditional Chinese medicine or Chinese patent medicine for infertility treatment in the last month(30 days).

Exit Criteria:

* subjects who have adverse events cannot be tolerated;
* severe breach of the protocol;
* for subjects who exit due to personal or unpredictable reasons, please describe specific details;
* subjects considered inappropriate to continue to participate in the study for other medical reasons.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1467 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongzi Yang, professor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (12):
- China (12):
  - Chongqing Health Center For Women and Children, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Liuzhou Maternal and Child Healthcare Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Reproductive and Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan
  - The Affiliated Suzhou Hospital of Nanjing Medical University, Suzhou, Jiangsu
  - Reproductive Hospital affiliated to Shandong University, Jinan, Shandong
  - Northwest Women and Children's Hospital, Xi’an, Shanxi
  - Tangdu Hospital of Air Force Medical University, Xi’an, Shanxi
  - West China Second University Hospital/West China Women's and Children's Hospital, Sichuan, Sichuan

REFERENCES:
- [Derived] Li Y, Gong F, Wang X, Hu L, Li H, Guan Y, Ye H, Fan L, Bai H, Wang Z, Huang W, Ma X, Yang D, Zhang H. Zishen Yutai Pill increased live births in advanced maternal age women: a randomized clinical trial. Nat Commun. 2025 Dec 24. doi: 10.1038/s41467-025-67714-4. Online ahead of print. PMID 41444477

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Started | 734 | 733
Completed | 419 | 409
Not Completed | 315 | 324

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zishen Yutai Pill Group | Placebo Group | Total
Number analyzed (Participants) | 734 | 733 | 1467
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.25 (1.80) | 37.25 (1.88) | 37.25 (1.84)
Age, Customized [Count of Participants; unit: Participants]
  Between 35 and 37 years | 425 | 426 | 851
  Between 38 and 39 years | 213 | 212 | 425
  Between 40 and 42 years | 96 | 95 | 191
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 734 | 733 | 1467
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 734 | 733 | 1467
Weight [Mean (Standard Deviation); unit: kilogram] | 57.79 (7.76) | 57.42 (7.51) | 57.61 (7.64)
Height [Mean (Standard Deviation); unit: centimeter] | 159.40 (5.38) | 159.14 (5.26) | 159.27 (5.32)
Type of infertility [Count of Participants; unit: Participants]
  Primary infertility | 181 | 171 | 352
  Secondary infertility | 545 | 554 | 1099
  Missing | 8 | 8 | 16
Duration of attempt to conceive [Median (Inter-Quartile Range); unit: years] | 3.0 [2.0 to 6.5] | 4.0 [2.0 to 7.0] | 4.0 [2.0 to 7.0]
Concomitant infertility factors [Number; unit: participants]
  Pelvic factors and tubal factors | 519 | 542 | 1061
  Endometriosis | 22 | 13 | 35
  Male factors | 331 | 345 | 676
  Unexplained factors | 35 | 25 | 60
  Ovulation disorder | 78 | 96 | 174
  Scar uterus | 88 | 93 | 181
  Obese/overweight | 69 | 75 | 144
  Diabetes | 32 | 35 | 67
Previous IVF cycle [Count of Participants; unit: Participants]
  0 | 604 | 591 | 1195
  1 | 54 | 71 | 125
  2 | 48 | 49 | 97
  ≥3 | 18 | 12 | 30
  Missing | 10 | 10 | 20
Previous miscarriage [Count of Participants; unit: Participants] | 138 | 148 | 286
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.72 (2.61) | 22.66 (2.64) | 22.69 (2.62)
Antral follicular count (AFC) [Median (Inter-Quartile Range); unit: Follicles] | 11 [7 to 16] | 11 [8 to 15] | 11 [7 to 16]
Anti-Müllerian hormone (AMH) [Median (Inter-Quartile Range); unit: ng/mL] | 2.10 [1.29 to 3.69] | 2.06 [1.16 to 3.36] | 2.09 [1.24 to 3.51]
Estradiol (E2) [Median (Inter-Quartile Range); unit: pmol/L] | 160.74 [113.99 to 238.21] | 159.61 [110.10 to 248.94] | 160.31 [112.67 to 244.17]
follicular-stimulating hormone (FSH) [Median (Inter-Quartile Range); unit: IU/L] | 6.83 [5.44 to 8.64] | 6.84 [5.31 to 8.49] | 6.83 [5.36 to 8.55]
Luteinizing hormone (LH) [Median (Inter-Quartile Range); unit: IU/L] | 4.05 [2.89 to 5.36] | 4.09 [3.01 to 5.50] | 4.08 [2.97 to 5.45]
Prolactin (PRL) [Median (Inter-Quartile Range); unit: mIU/L] | 281.85 [207.81 to 384.67] | 283.66 [198.75 to 387.91] | 282.17 [202.73 to 389.74]
Testerone (T) [Median (Inter-Quartile Range); unit: nmol/L] | 0.90 [0.59 to 1.37] | 0.94 [0.59 to 1.38] | 0.90 [0.59 to 1.38]

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate
Description: Live birth rate=Number of live birth / Paticipants randomized
Time Frame: 1 year after embryo transfer day, up to a maximum duration of 58 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
Participants | 171 | 139
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.042, Chi-squared; Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.01 to 1.50]

2. Secondary Outcome: Number of Retrieved Oocytes
Description: The total number of oocytes retrieved through ultrasound-guided transvaginal aspiration.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: oocytes
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
oocytes | 9 [5 to 13] | 9 [6 to 13]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.781, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rate of Retrieved Oocytes
Description: Rate of retrieved oocytes =Number of retrieved oocytes/Number of follicles with a diameter ≥10mm on the HCG injection day.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: percentage of retrieved oocytes
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
percentage of retrieved oocytes | 85.7 [68.3 to 109.1] | 88.9 [69.2 to 107.9]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.609, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Matured Oocytes Retrieved
Description: The number of oocytes with pronuclei or polar bodies observed on Day 1 after oocyte retrieval in IVF patients, or as the number of MII oocytes on the day of oocyte retrieval in ICSI patients.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: oocytes
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
oocytes | 8 [5 to 11] | 7 [4 to 11]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.528, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rate of Matured Oocytes
Description: Rate of mature oocytes = Number of mature oocytes/Number of retrieved oocytes
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: percentage of matured oocytes
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
percentage of matured oocytes | 90.0 [77.8 to 100.0] | 90.9 [77.7 to 100.0]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.880, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Cleavage
Description: Number of fertilized oocytes that undergo cleavage on Day 2 after oocyte retrieval.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: oocytes
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
oocytes | 7 [4 to 10] | 6 [4 to 10]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.289, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Cleavage Rate
Description: Cleavage rate=Number of all cleaved embryos/Number of fertilized oocytes (2PN+1PN+ multiple PN)
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: percentage of cleaved embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
percentage of cleaved embryos | 91.0 [70.0 to 100.0] | 90.0 [71.4 to 100.0]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.860, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Available Embryos
Description: The sum of the number of embryos transferred and the number of embryos frozen.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
embryos | 4 [2 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.163, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Rate of Available Embryos
Description: Rate of available embryos=Number of available embryos/Number of cleaved oocytes.
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: percentage of available embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
percentage of available embryos | 57.1 [40.0 to 75.0] | 50.0 [37.8 to 71.4]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.197, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of High-quality Embryos
Description: High-quality embryo will be defined according to the day of embryo transfer, following the Istanbul consensus and Gardner criteria, Day 2: 4 cells, cell fragments <10% and no multi-nucleus; Day 3: 8 cells, cell fragments <10%, no multi-nucleus; Day 5: stage 4 blastocyst, grade A inner cell mass, grade A trophectoderm (12,13).
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
embryos | 2 [0 to 4] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.178, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Rate of High-quality Embryos
Description: Rate of high-quality embryos=Number of high-quality embryos/Number of available embryos
Time Frame: On embryo transfer day, approximately 6 weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: percentage of high-quality embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
percentage of high-quality embryos | 50.0 [0.0 to 100.0] | 50.0 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.549, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Biochemical Pregnancy Rate
Description: Biochemical pregnancy rate=Number of positive pregnancy tests/Paticipants randomized
Time Frame: 14 days after ET day, approximately 8 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
Participants | 232 | 195
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.035, Chi-squared; Risk Ratio (RR) = 1.19, 95% CI 2-sided [1.01 to 1.40]

13. Secondary Outcome: Implantation Rate
Description: Implantation rate=Number of gestational sacs/Number of embryos transferred
Time Frame: five weeks after ET day, approximately 11 weeks
Population: Number of embryos transferred
Measure: Count of Units; unit: embryos
Units Other Than Participants: embryos
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 422 | 412
Number analyzed (embryos) | 700 | 667
embryos | 252 | 204
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.034, Chi-squared; Risk Ratio (RR) = 1.18, 95% CI 2-sided [1.01 to 1.37]

14. Secondary Outcome: Clinical Pregnancy Rate
Description: The clinical pregnancy determined by the ultrasound, and Clinical pregnancy rate=Number of clinical pregnancies / Paticipants randomized
Time Frame: five weeks after ET day, approximately 11 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 734 | 733
Participants | 216 | 177
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.022, Chi-squared; Risk Ratio (RR) = 1.22, 95% CI 2-sided [1.03 to 1.45]

15. Secondary Outcome: Miscarriage Rate (Among Positive Pregnancy Test Population)
Description: Miscarriage Rate (among positive pregnancy test population) =Number of miscarriages / Number of biochemical pregnancy
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: Population with serum β-HCG positive during pregnancy tests
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 232 | 195
Participants | 57 | 51
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.707, Chi-squared; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.68 to 1.30]

16. Secondary Outcome: Miscarriage Rate (Among Clinical Pregnancy Population)
Description: Miscarriage rate (among clinical pregnancy population)=Number of miscarriages / Number of clinical pregnancies
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: Population with intrauterine gestation sac with fetal motion under transvaginal ultrasonography
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 216 | 177
Participants | 45 | 38
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.878, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.66 to 1.42]

17. Secondary Outcome: The Birth Weight of the Newborn
Description: By checking medical records
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: Newborns (145 singletons and 26 pairs of twins in Zishen Yutai pill group, 117 singletons and 22 pairs of twins in placebo group)
Measure: Median (Inter-Quartile Range); unit: gram
Units Other Than Participants: Neonates
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Number analyzed (Neonates) | 197 | 161
gram
  Singleton: number analyzed (Participants) | 145 | 117
  Singleton: number analyzed (Neonates) | 145 | 117
  Singleton | 3250.0 [2972.5 to 3542.5] | 3260.0 [3000.0 to 3600.0]
  Twin: number analyzed (Participants) | 26 | 22
  Twin: number analyzed (Neonates) | 52 | 44
  Twin | 2450.0 [2150.0 to 2600.0] | 2275.0 [2085.0 to 2595.0]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Singleton; Test type: Other; p = 0.564, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Zishen Yutai Pill Group vs Placebo Group; Twin; Test type: Other; p = 0.417, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: The Birth Height of the Newborn
Description: By checking medical records
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: centimeter
Units Other Than Participants: Neonates
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Number analyzed (Neonates) | 197 | 161
centimeter
  Singleton: number analyzed (Participants) | 145 | 117
  Singleton: number analyzed (Neonates) | 145 | 117
  Singleton | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Twin: number analyzed (Participants) | 26 | 22
  Twin: number analyzed (Neonates) | 52 | 44
  Twin | 48.0 [47.0 to 49.0] | 48.0 [45.0 to 49.0]
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Singleton; Test type: Other; p = 0.985, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Zishen Yutai Pill Group vs Placebo Group; Twin; Test type: Other; p = 0.157, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Preterm Delivery Among Live Birth
Description: Delivery of a fetus at less than 37 and more than 28 weeks gestational age.
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: Participants who had live birth
Measure: Count of Participants; unit: Participants
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Participants | 29 | 22
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.789, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.65 to 1.78]

20. Secondary Outcome: Low Birth Weight Among Neonates
Description: Neonatal birth weight ≤ 2500 g.
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: as for outcome 17
Measure: Count of Units; unit: Neonates
Units Other Than Participants: Neonates
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Number analyzed (Neonates) | 197 | 161
Neonates | 24 | 18
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.769, Chi-squared; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.61 to 1.94]

21. Secondary Outcome: Congenital Anomalies Among Neonates
Description: Congenital anomalies are defined as structural or functional anomalies that occur during intrauterine life, including minor and major anomalies.
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: as for outcome 17
Measure: Count of Units; unit: neonates
Units Other Than Participants: neonates
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Number analyzed (neonates) | 197 | 161
neonates | 1 | 2
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.590, Fisher Exact; Risk Ratio (RR) = 0.41, 95% CI 2-sided [0.04 to 4.45]

22. Secondary Outcome: Neonates Entering NICU
Description: NICU, neonate intensive care unit.
Time Frame: 1 year after embryo transfer, up to 58 weeks
Population: as for outcome 17
Measure: Count of Units; unit: neonates
Units Other Than Participants: neonates
Arm/Group | Zishen Yutai Pill Group | Placebo Group
Number analyzed (Participants) | 171 | 139
Number analyzed (neonates) | 197 | 161
neonates | 5 | 2
Statistical Analysis 1: Comparison: Zishen Yutai Pill Group vs Placebo Group; Test type: Other; p = 0.465, Fisher Exact; Risk Ratio (RR) = 2.04, 95% CI 2-sided [0.40 to 10.39]

ADVERSE EVENTS:
Time Frame: From enrollment until 1 year after ET, up to 58 weeks
Description: maternal and neonatal adverse events
Arm/Group | Zishen Yutai Pill Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/734 | 0/733
Serious Adverse Events (participants affected / at risk) | 22/734 | 18/733
Other Adverse Events (participants affected / at risk) | 0/734 | 0/733
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Zishen Yutai Pill Group (N=734) | Placebo Group (N=733)
Ovarian hyperstimulation syndrome (Endocrine disorders) | 4 (4) | 6 (6) — Moderate to severe ovarian hyperstimulation syndrome
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 12/232 (12) | 7/195 (7) — Hospitalization due to miscarriage
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 4/232 (4) | 5/195 (5)
Cryptorchidism (Congenital, familial and genetic disorders) | 1/197 (1) | 0/161 (0) — Neonatal congenital cryptorchidism
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Congenital atrial septal defect (Congenital, familial and genetic disorders) | 1/197 (1) | 0/161 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03703700/Prot_SAP_000.pdf